CLINICAL TRIAL: NCT02474615
Title: Applicability Clinic of Cement Portland Structural White in Endodontic Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Sergio Ribeiro da Silva, Aplicability clinic of cement Portland structural additived white in surgery paraendodontic, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14099
Record Dates: First submitted 2015-02-24; First posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Mandibular Hypoplasia
Keywords: Apicoectomy; Oral surgery; Biocompatible materials; Dental Cements; Translational Medical Research
MeSH Terms: conditions — Micrognathism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TOOTH ENDODONTIC SURGERY - PBEA (Experimental): Endodontic surgery 15 teeth - PBEA
  Interventions: Procedure: ENDODONTIC SURGERY
- TOOTH ENDODONTIC SURGERY -MTA (Experimental): Endodontic surgery 15 teeth - MTA
  Interventions: Procedure: ENDODONTIC SURGERY

INTERVENTIONS:
Procedure: ENDODONTIC SURGERY — ENDODONTIC SURGERY

SUMMARY:
Thirty teeth twelve patients, two female and a male, who had persistent periradicular lesions were selected to participate in this study. The lesions were diagnosed with cone-beam computed tomography (cone-beam CT; Model i-Cat 17-19, Imaging Sciences International LLC).In patients with two teeth to be treated, a tooth was retroobturado with PBEA cement, (experiment) and another tooth was retroobturado with MTA cement (control).

There was significance for the two cements on the repair of wounds. Key words: Apicoectomy; Oral Surgery; Biocompatible Materials; Dental Cements; Translational Medical Research

DETAILED DESCRIPTION:
Objective: to evaluate the clinical applicability of structural Portland white cement additive in retrofilling surgeries. Method: persistent apical periodontitis 30 teeth of 12 patients were diagnosed by computed tomography CT, cone beam. Each of them had from two to four compromised teeth. The endodontic surgery were performed and the teeth were retrofilling Each patient had a retrofilling tooth with cement mineral trioxide aggregate (MTA) control and other tooth with white Portland cement structural additive (PBEA) experiment. When the patient presented four teeth with injury, two were retrofilling with MTA and two Portland cement with structural white cement additive. Six months after surgery, there were new scans to evaluate the repair or not the wounds.

ELIGIBILITY:
Inclusion Criteria:

* patients were diagnosed by computed tomography CT, cone beam
* each of them had from two to four compromised teeth

Exclusion Criteria:

* patients who did not return for review after six months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Regeneration measured by tomographers endodontic surgery | Six months after surgery
  Six months after surgery, there were new scans to evaluate the repair or not the wounds.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Francescato Veiga, Study Director — BRAZIL, UNIVAS

REFERENCES:
- [Background] da Silva SR, da Silva Neto JD, Veiga DF, Schnaider TB, Ferreira LM. Portland cement versus MTA as a root-end filling material. A pilot study. Acta Cir Bras. 2015 Feb;30(2):160-4. doi: 10.1590/S0102-865020150020000011. PMID 25714696
- [Result] Silva Neto JD, Schnaider TB, Gragnani A, Paiva AP, Novo NF, Ferreira LM. Portland cement with additives in the repair of furcation perforations in dogs. Acta Cir Bras. 2012 Nov;27(11):809-14. doi: 10.1590/s0102-86502012001100011. PMID 23117614
- [Result] Feldman AM. Does academic culture support translational research? Clin Transl Sci. 2008 Sep;1(2):87-8. doi: 10.1111/j.1752-8062.2008.00046.x. No abstract available. PMID 20443823
- [Result] Silva Neto JD, Brito RH, Schnaider TB, Gragnani A, Engelman M, Ferreira LM. Root perforations treatment using mineral trioxide aggregate and Portland cements. Acta Cir Bras. 2010 Dec;25(6):479-84. doi: 10.1590/s0102-86502010000600004. PMID 21120277